CLINICAL TRIAL: NCT04814732
Title: An Expanded Access Program of Surufatinib for Patients With Advanced or Metastatic Neuroendocrine Tumors
Brief Title: Expanded Access Program of Surufatinib
Status: No longer available | Type: Expanded Access
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-012-GLOB3
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Surufatinib — HMP-012

SUMMARY:
This treatment protocol is intended to provide early access of surufatinib to patients with locally advanced or metastatic NETs for whom, in the opinion of their treating physician, other treatment options or surufatinib clinical trials in this indication are unsuitable. This EAP is currently available in the US only.

DETAILED DESCRIPTION:
Prior to any assessments, all subjects must provide a signed ICF. Prior to inclusion in the program, the patients must undergo all appropriate screening procedures to check for eligibility.

Once eligibility is confirmed, patients will receive treatment with surufatinib 300mg, orally (PO), daily (QD). All patients will undergo continuous monitoring for safety until the end of treatment.

There is no pre-defined duration of treatment for each patient. Patients will be treated until progressive disease (as defined by treating physician), unacceptable toxicity, death, withdrawal from program, the treatment becomes commercially available, or halting of product development.

A follow-up clinic visit is recommended for all patients approximately 30 days after last dose of treatment to complete the final safety assessments, as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented, well differentiated, locally advanced or metastatic NETs
2. The patient or parent/legal guardian (as appropriate) is willing and able to provide informed consent, and where required, the patient is willing to provide assent
3. ≥12 years of age
4. In the opinion of the patient's treating physician, other treatment options or clinical trials in this indication are unsuitable
5. Patient has adequate bone marrow and organ function
6. Urine dipstick ≤1+ for proteinuria or ≤30 mg/dL in urinalysis,
7. ECOG ≤2 for adult patients (≥18 years of age), Karnofsky ≥60 for patients >16 and <18 years of age, and Lansky ≥60 for pediatric patients ≤16 years of age
8. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and partner) to use a highly effective form(s) of contraception

Exclusion Criteria:

1. Uncontrollable hypertension, as defined by local institution
2. Gastrointestinal disease or condition that the physician suspects may affect drug absorption
3. History or presence of a serious hemorrhage
4. Clinically significant cardiovascular disease
5. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy
6. High risk of bleeding at screening due to tumor invasion
7. Arterial thrombosis or deep venous thrombosis within 6 months prior to first dosing or thromboembolic events (including stroke and/or transient ischemic attack) within 6 months prior to first dosing
8. Received treatment with anticancer therapy, including investigational therapy, within 7 days or 5 half-lives (whichever is longer)
9. Received prior treatment with surufatinib
10. Inability to take medication orally
11. Any other clinically significant comorbidities that, in the judgment of the treating physician, could predispose the patient to safety risks

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Hahka-Kemppinen, MD, Study Chair — Hutchison Medipharma Limited
Locations (11):
- United States (11):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Mercy Medical Center, Medical Oncology & Hematology, Baltimore, Maryland
  - Karmanos Cancer Center, Detroit, Michigan
  - MidAmerica Cancer Care, Kansas City, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Providence Cancer Institute Franz Clinic, Providence Health & Services, Portland, Oregon
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Intermountain Healthcare, Murray, Utah
  - Intermountain Cancer Center, St. George, Utah